CLINICAL TRIAL: NCT05508178
Title: A Phase 1 Randomised, Double-Blind, Placebo-Controlled, Safety and Immunogenicity Study of a Plant-Produced, Bivalent, Recombinant Norovirus-Like Particle Vaccine, Administered Intramuscularly to Healthy Adults Aged 18 to 40 Years
Brief Title: Recombinant, Bivalent, Norovirus Vaccine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icon Genetics GmbH (Industry)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: rNV-2v-001
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Norovirus
Keywords: Norovirus; Vaccine; Adults; Safety; Immunogenicity; First-in-human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (100 µg) (Experimental): Participants 18-40 years of age, 2-dose regimen: Norovirus bivalent GI.4 (50 μg) / GII.4 (50 μg) virus-like particle (VLP) vaccine, intramuscularly (IM), on Day 1 and Day 29
  Interventions: Biological: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (100 µg)
- Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (300 µg) (Experimental): Participants 18-40 years of age, 2-dose regimen: Norovirus bivalent GI.4 (150 μg) / GII.4 (150 μg) virus-like particle (VLP) vaccine, intramuscularly (IM), on Day 1 and Day 29
  Interventions: Biological: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (300 µg)
- Placebo (Placebo Comparator): Participants 18-40 years of age, 2-dose regimen: Placebo (norovirus vaccine vehicle without antigens), intramuscularly (IM), on Day 1 and Day 29
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (100 µg) — Norovirus: 50 µg GI.4 VLP + 50 µg GII.4 VLP without adjuvant
  Other Names: rNV-2v
  Arms: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (100 µg)
Biological: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (300 µg) — Norovirus: 150 µg GI.4 VLP + 150 µg GII.4 VLP without adjuvant
  Other Names: rNV-2v
  Arms: Norovirus GI.4 / GII.4 Bivalent VLP Vaccine (300 µg)
Drug: Placebo — Norovirus vaccine (rNV-2v) vehicle without antigen
  Other Names: Vehicle
  Arms: Placebo

SUMMARY:
This clinical study will evaluate the vaccine candidate rNV-2v, which is under development to prevent disease triggered by noroviruses. Noroviruses are one of the leading causes of gastrointestinal diseases in the world. Norovirus infections can cause vomiting, diarrhea, and cramping. Noroviruses can spread easily, especially in hospitals, schools, military barracks and ships. At the moment, there is no vaccine available to prevent norovirus infections or disease. This clinical trial will look at the safety and tolerability of an investigational vaccine that is being developed to prevent norovirus-related disease. The trial will also look at whether the immune system produces a response to the investigational study vaccine. The study vaccine is a combination of two different types of norovirus antigens. In contrast to similar vaccines under development, the vaccine studied here adds no substances (adjuvants) to increase or modulate the immune response. The study vaccine is produced using a plant-based system rather than a typically used animal cell system. This is the first time the study vaccine will be given to humans. Two different doses of the investigational study vaccine will be tested in this trial. Either the investigational study vaccine or the placebo will be given as 2 injections. These injections will be given about 1 month apart. The trial will last about 12 months, from the time of enrollment.

DETAILED DESCRIPTION:
The vaccine being tested in this study is rNV-2v; norovirus GI.4/GII.4 bivalent, virus-like particle (VLP) vaccine without adjuvant. Two norovirus vaccine dose levels (50 µg + 50 µg and 150 µg + 150 µg) are being tested for safety, tolerability and immunogenicity in a young adult population (18-40 years of age).

The study will enroll 60 participants. Participants will be randomly assigned to one of three treatment groups.

Norovirus GI.4/GII.4 bivalent VLP vaccine (50 µg + 50 µg), 2 administrations Norovirus GI.1/GII.4 bivalent VLP vaccine (150 µg + 150 µg), 2 administrations Placebo (norovirus vaccine vehicle without antigens), 2 administrations All participants randomized will be administered either norovirus vaccine or placebo on Day 1 and on Day 29 of the study.

Participants will be asked to record any reactions/ symptoms that may be related or not to the vaccine in a diary card for 7 days after each vaccination. Unsolicited Adverse Events (AEs) will be recorded through open-ended inquiries for 28 days after each vaccine administration. Serious AEs will be captured until Day 365.

This single-center trial will be conducted at the Center for Vaccinology (CEVAC), Ghent, Belgium. Participants will make multiple visits to the clinic including a final visit on Day 365.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Male or female aged 18 to 40 years (inclusive) at Screening.
3. Good general health as determined by a Screening evaluation that includes vital signs, medical history, physical examinations, and laboratory assessments within 28 days before administration of the study vaccine.
4. Expressed interest, availability and understanding to fulfil the study requirements, and in the opinion of the Investigator, can and will comply with the protocol requirements.
5. Female subjects of childbearing potential must be using a highly-effective licensed method of birth control for 30 days prior to the first vaccination and must agree to continue such precautions during the study until 60 days after the second vaccination. Male subjects must agree to employ barrier contraception from the day of first vaccination until 60 days after the second vaccination, if their female partner of childbearing potential doesn't use a highly effective method of birth control.
6. Agrees not to participate in another clinical study with an investigational product or to use any nonregistered product (drug, vaccine, or medical device) for the duration of the study.

Exclusion Criteria:

Any condition that may interfere with study participation or place the participant at increased risk of AEs would be excluded from the study. Additionally, subjects are excluded from the study if any of the following criteria apply:

1. Positive serology test results for hepatitis C virus, human immunodeficiency virus antibody, and/or hepatitis B surface antigen at Screening.
2. Pregnant or lactating women.
3. History of any of the following medical illnesses, which, in the opinion of the Investigator, may interfere with study participation or place the participant at increased risk of AEs, including but not limited to: immunosuppression (disease or treatments that may affect immune system function), diabetes, cancer (malignancy other than a resolved or excised skin lesion), heart disease (hospitalisation for a heart attack, arrhythmia, or syncope), unconsciousness (excluding single and brief concussion), seizures, asthma requiring treatment with inhaler or medication in the past 2 years, neuroinflammatory disease, autoimmune disease, recurrent infections (more than 3 hospitalisations for invasive bacterial infections such as pneumonia or meningitis).
4. Any current or chronic conditions requiring daily medication other than vitamins, minerals, or antihypertensives, as per the Investigator's discretion. Rescreening for acute illness that is expected to resolve quickly is allowed, as per the Investigator's discretion.
5. Known or suspected allergies or hypersensitivity to any component of the study vaccine.
6. Any clinically significant abnormality detected during physical examinations or vital sign evaluations, as per the Investigator's discretion.
7. Hypertension defined as a mean of triplicate sitting blood pressure measurements >150/90 mmHg.
8. Any Screening hematology or biochemistry abnormalities considered clinically significant by the Investigator.
9. For women of child bearing potential, positive urine/serum pregnancy test at Screening or within 24 hours of the first dose of the study vaccine.
10. Body (oral) temperature >38°C or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days of administration of the first dose of the study vaccine.
11. Administration of rNV-2v or any other experimental norovirus vaccine in the past.
12. Planned administration of other vaccines from 14 days before the first administration of the study vaccine and 60 days after the last study administration of the study vaccine, with the exception of inactivated influenza vaccine, which can be administered up to 14 days before or from 30 days after the last administration of the study vaccine.
13. Administration of immunoglobins or any blood products within 180 days prior to the first administration of the study vaccine and throughout the study duration, as per the Investigator's discretion.
14. Relatives of the Sponsor, clinical research organisation, or the study centre personnel are excluded from participating in the study.
15. History of psychiatric hospitalisation, alcohol abuse, or illicit drug use, which in the opinion of the Investigator, may affect the subject's participation in the study.
16. Other condition that in the clinical judgement of the Investigator would jeopardise the safety or rights of a subject participating in the study, would render the subject unable to comply with the protocol, or would interfere with the evaluation of the study vaccine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
To assess the safety, tolerability, and reactogenicity of rNV-2v administered intramuscularly (IM) to healthy subjects | within 7 days after each administration of the vaccine
  Safety and tolerability as determined by:
  * The occurrence of adverse events (AEs) consisting of local and systemic signs and symptoms within 7 days after vaccination. Local and systemic signs and symptoms, assessed as typical and expected reactions to study vaccine administration including pain, redness, and swelling at the injection site; fever, fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhea, and/or abdominal pain), headache, myalgia, shivering, and arthralgia.
  * Incidence of abnormal hematology and serum chemistry laboratory values.
  * Occurrence of serious adverse events (SAEs).
  * Onset of any significant new medical conditions following the first administration of study vaccine.
To assess the safety, tolerability, and reactogenicity of rNV-2v administered intramuscularly (IM) to healthy subjects | until 28 days after second administration of study vaccine (Day 57)
  Safety and tolerability as determined by:
  * Incidence of abnormal hematology and serum chemistry laboratory values.
  * Occurrence of serious adverse events (SAEs).
  * Onset of any significant new medical conditions following the first administration of study vaccine.
To assess the safety, tolerability, and reactogenicity of rNV-2v administered intramuscularly (IM) to healthy subjects | for 364 days following the first administration of study vaccine
  Safety and tolerability as determined by:
  * Occurrence of serious adverse events (SAEs).
  * Onset of any significant new medical conditions following the first administration of study vaccine.

SECONDARY OUTCOMES:
To assess the humoral immune response elicited by rNV-2v by measuring binding antibodies against the GI.4 and GII.4 components of the bivalent vaccine | Pre-dose, Week 1, Week 4, Week 8, Week 26, and Week 52.
  virus-like particle (VLP) antigens, relative to Baseline:
  - Anti-GI.4 and GII.4 VLP immunoglobulin (Ig) G titer by enzyme-linked immunosorbent assay (ELISA) in serum

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Center for Vaccinology (CEVAC), Ghent University and University Hospital, Ghent, Belgium.
Locations (1):
- Center for Vaccinology (CEVAC), Ghent University and University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waerlop G, Janssens Y, Jacobs B, Jarczowski F, Diessner A, Leroux-Roels G, Klimyuk V, Leroux-Roels I, Thieme F. Immune responses in healthy adults elicited by a bivalent norovirus vaccine candidate composed of GI.4 and GII.4 VLPs without adjuvant. Front Immunol. 2023 Jun 26;14:1188431. doi: 10.3389/fimmu.2023.1188431. eCollection 2023. PMID 37435073
- [Derived] Leroux-Roels I, Maes C, Joye J, Jacobs B, Jarczowski F, Diessner A, Janssens Y, Waerlop G, Tamminen K, Heinimaki S, Blazevic V, Leroux-Roels G, Klimyuk V, Adachi H, Hiruta K, Thieme F. A randomized, double-blind, placebo-controlled, dose-escalating phase I trial to evaluate safety and immunogenicity of a plant-produced, bivalent, recombinant norovirus-like particle vaccine. Front Immunol. 2022 Oct 7;13:1021500. doi: 10.3389/fimmu.2022.1021500. eCollection 2022. PMID 36275772
- See also: Center for Disease Control and Prevention norovirus information webpage — https://www.cdc.gov/norovirus/index.html